CLINICAL TRIAL: NCT05847179
Title: A Phase 2, Open-Label Study to Evaluate the Safety and Tolerability of Progerinin for the Treatment of Bone Mineral Density (BMD) Loss in Subjects With Typical Werner Syndrome
Brief Title: Phase 2, Open-Label Study to Evaluate the Safety and Tolerability of Progerinin in Werner Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PRG Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG-PRO-004
Record Dates: First submitted 2023-03-31; First posted 2023-05-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Werner Syndrome
MeSH Terms: conditions — Werner Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): all subjects will receive Progerinin 2400mg (1200mg twice daily) after morning and evening meals for a year
  Interventions: Drug: Progerinin

INTERVENTIONS:
Drug: Progerinin — This is a Phase 2, open-label study to evaluate the safety and Tolerability of Progerinin for the treatment of BMD Bone Mineral Density (BMD) Loss in Subjects with Typical Werner Syndrome.
  . There will be up to 5 subjects that will receive treatment with Progerinin twice daily for approximately 1 year. This study will have three phases: Screening Phase, Treatment Phase, and Follow-Up Phase.

SUMMARY:
This is a Phase 2, open-label study to A Phase 2, Open-Label Study to Evaluate the Safety and Tolerability of Progerinin for the Treatment of Bone Mineral Density (BMD) Loss in Subjects with Typical Werner Syndrome.

There will be up to 5 subjects that will receive treatment with Progerinin twice daily for approximately 1 year.

DETAILED DESCRIPTION:
Subjects who have successfully completed the Screening phase will enter the baseline and treatment phase of the study. Subjects will take the assigned treatment of Progerinin (2400 mg) split as 1200 mg BID in the morning and evening with food for 1-Year.

To evaluate the safety and tolerability of Progerinin for the treatment of BMD loss in subjects with typical Werner syndrome.

The secondary objectives of this study are:

* To characterize the activity of Progerinin on bone metabolism in subjects with typical Werner syndrome.
* To evaluate the pharmacokinetics (PK) of Progerinin sachet administered twice daily (BID) in subjects with typical Werner syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least ≥ 18 years of age.
2. Subjects should have a confirmed diagnosis of typical Werner syndrome by genetic analysis.
3. Subjects should be osteopenic (T-score between -1.0 and -2.5) or have confirmed osteoporosis (Tscore ≤ -2.5) at screening/baseline. Subjects may continue to receive bone supplements (e.g., bisphosphonates, calcium supplements, Vitamin D supplements, etc.) as appropriate per standard of care throughout the study.
4. Male or non-pregnant, non-lactating female.
5. Subjects screening blood chemistry inclusive of metabolic panel, hematology, and urine analysis results should be acceptable to the investigator.
6. Negative pregnancy test for female subjects as described below. Women of child bearing potential (WOCBP) and Women not of child-bearing potential are eligible to participate. Both women of childbearing potential and women of non-child-bearing potential should use an approved method of birth control and agrees to continue to use this method for the duration of the study and for 90 days after last treatment.

   Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, implanted, or injected) in conjunction with a barrier method (WOCBP only), female subject/partner's use of an intrauterine device (IUD), or if the female subject/partner is surgically sterile or two years post-menopausal. All male subjects/partners must agree to use a In addition, subjects may not donate sperm for the duration of the study and for 90 days after last treatment.

   Females who are less than two (2) years post-menopausal, those with tubal ligations and those using contraception must have a negative serum pregnancy test at baseline within the one (1) week prior to the first study medication administration. Every six weeks, and at study termination a pregnancy test should be performed, either serum or urine stick test. However, if the urine result is positive, a serum pregnancy test will be performed.
7. Provide signed written informed consent and willingness, ability to comply with study requirements.
8. Subject must have a projected life expectancy of ≥ 12 months in the opinion of the Investigator.

Exclusion Criteria:

1. Subject with clinical signs seen at screening are at the final stage of Werner syndrome progression, and completion of the study is difficult to be assessed, including:

   * Subjects who received continuous or intermittent home oxygen therapy for 6 months before obtaining consent
   * Subjects who received at least 2 hospitalizations for pneumonia during the 12 months prior to obtaining consent
   * Subjects who have at least 10% net weight loss and have not recovered. This includes significant net weight loss over the last six months.
2. Subjects with significant dehydration as judged by the principal investigator.
3. Subjects with pericardial fluid, ascites and pleural effusion.
4. Therapy with investigational drugs within 30 days of beginning study medication.
5. History of prior malignancy, except for adequately treated in situ cancer, basal cell, squamous cell skin cancer, or other cancers (e.g., breast, prostate) for which the subject has been disease-free for at least 3 years.
6. Any serious medical condition, laboratory abnormality, psychiatric illness, or comorbidity that, in the judgment of the Investigator, would make the subject inappropriate for the study.
7. Serious systemic fungal, bacterial, viral, or other infection that is not controlled or requires intravenous (IV) treatment for infection(s).
8. Subjects with known history of having Acquired Immunodeficiency Syndrome (AIDS) or with a history known to be infected with Human Immunodeficiency Virus (HIV).
9. Subjects with a history of serious drug hypersensitivity or allergic reaction such as anaphylaxis or any component of the formulation.
10. Clinically significant bleeding within 2 weeks prior to baseline (e.g., gastrointestinal [GI] bleeding, intracranial hemorrhage).
11. Medical or recreational use of marijuana or THC-containing compounds within 3 months of screening visit and for the duration of the trial.
12. Pregnant or lactating women.
13. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e., larger than what is required for placement of central venous access, percutaneous feeding tube, or biopsy), within 28 days prior to baseline or anticipated surgery during the study period.
14. Inability to return for scheduled treatment and assessments.
15. Subjects that require concomitant use of any medications or substances that are strong inhibitors or inducers of CYP2D6 or CYP2C8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events (TEAEs) | week 54
  The intensity of the event will be graded using CTCAE v5.0 criteria
Incidence of Treatment-Related Adverse Events | week 54
Incidence of Serious Adverse Events (SAEs) | week 54
Incidence of TEAEs and SAEs leading to discontinuation of study medication | week 54
Changes in Blood Hemoglobin (g/dl) from baseline | week 54
Changes in Blood White Blood Cell (cell per microliter) from baseline | week 54
Changes in Blood Platelets (cell per microliter) from baseline | week 54
Changes in Serum Creatinine (µmol/L) from baseline | week 54
Changes in Serum Alanine Aminotransferase (IU/l) from baseline | week 54
Changes in Serum Aspartate Aminotransferase (IU/l) from baseline | week 54
Changes in Serum Alkaline Phosphatase (microkatal per liter) from baseline | week 54
Changes in weight (kg) from baseline | week 54
Changes in pulse rate (beats per minute) from baseline | week 54
Changes in respiratory rate (breaths per minute) from baseline | week 54
Changes in temperature (°F) from baseline | week 54
Changes in systolic Blood pressure (mm Hg) from baseline | week 54
Changes in Diastolic Blood pressure (mm Hg) from baseline | week 54
Change in ECG ventricular rate from baseline (beats per minute) | week 54
Change in ECG PR interval (msec) | week 54
Change in ECG QRS interval (msec) | week 54
Change in ECG QT interval (msec) | week 54
Change in ECG QTc interval (msec) | week 54